CLINICAL TRIAL: NCT03992742
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2019: Personalized Cocktail Interventions to Increase Abstinence: a Sequential, Multiple Assignment, Randomized Trial (SMART)
Brief Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW 2019
Record Dates: First submitted 2019-06-12; First posted 2019-06-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Quit to Win; Cocktail intervention; SMART design
MeSH Terms: conditions — Smoking Cessation | interventions — corticosteroid hormone-induced factor; Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (subgroup A+B+C) (Experimental): Personalized instant messaging (PIM) + optional cocktail interventions (OCI) + AWARD advice + referral card + warning leaflet+ COSH booklet
  Interventions: Behavioral: Initial phase: personalized instant messaging (PIM); Behavioral: Second phase: optional cocktail interventions (OCI); Behavioral: AWARD advice; Behavioral: Warning leaflet; Behavioral: Referral card; Behavioral: COSH booklet
- Control Group (subgroup D+E+F) (Experimental): Regular instant messaging (RIM) + personalized instant messaging (PIM) + AWARD advice + referral card + warning leaflet+ COSH booklet
  Interventions: Behavioral: Initial phase: regular instant messaging (RIM); Behavioral: Second phase: personalized instant messaging (PIM); Behavioral: AWARD advice; Behavioral: Warning leaflet; Behavioral: Referral card; Behavioral: COSH booklet

INTERVENTIONS:
Behavioral: Initial phase: personalized instant messaging (PIM) — intervention Group participants will receive three months of personalized interaction through IM Apps (e.g. WhatsApp, WeChat). Our counsellors will trigger the conversation and encourage the participants to set a quit day. A total of pre-set 26 messages will be sent with the schedule of once daily for 1 week (the week across the quit date), 3 times a week for 4 weeks (2 weeks each before and after the week with quit date) and once a week for remaining 7 weeks. These messages covered generic information about the benefits of quitting, methods to avoid/ manage craving or withdrawal symptoms, and encouragement to quit and use SC services.
  At the end of the initial phase (1-month), complete responders (quitters) will continue to receive PIM (subgroup C). Incomplete responders (smokers) will be randomized to continue PIM (subgroup B) or receive OCI (subgroup A).
  Arms: Intervention Group (subgroup A+B+C)
Behavioral: Second phase: optional cocktail interventions (OCI) — For incomplete respondents (subgroup A) randomized to OCI, the available intervention options include multi-media messages, active referral plus financial incentive, phone counseling, family/peer support and medications (NRT). Participants will be guided by cessation counsellors at 1-month follow-up telephone survey to choose any combination of OCI based on their preference. If OCI participants cannot be followed up at 1-month, they will receive multi-media messages by default.
  Arms: Intervention Group (subgroup A+B+C)
Behavioral: Initial phase: regular instant messaging (RIM) — Participants enrolled in the Control Group will receive regular messages via IM services (e.g. WhatsApp, WeChat) since initial contact and until 3-month after baseline with a tapering schedule: 1) Baseline to 4-week (1-month): 2 times/ week (8 in total); 2) 4-week to 12-week (2- & 3-month): 1 time/week (8 in total).
  SC messages will generally include benefits of SC, encouragement on abstinence and use of SC services, tips on avoiding/ handling craving and reminder of participating in telephone follow-up. A reminder to participate in the telephone follow-up will also be sent at 1-, 2-, 3- and 6-month, making up a total of 20 messages.
  At the end of the initial phase (1-month), complete responders (quitters) will continue to receive RIM (subgroup F). Incomplete responders (smokers) will be second randomized to continue RIM (subgroup E) or receive PIM (subgroup D). Those who are unable to follow up at 1-month will be considered as nonresponsive to the intervention.
  Arms: Control Group (subgroup D+E+F)
Behavioral: Second phase: personalized instant messaging (PIM) — For incomplete responders allocated to PIM (subgroup D), participants will receive the same intervention as the Group A delivered at the initial stage. Participants will receive two months of personalized interaction through IM application. Please refer to Intervention Group "Initial phase: personalized instant messaging (PIM)" for details.
  Arms: Control Group (subgroup D+E+F)
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date).
  Other Names: Ask, Warn, Advise, Refer, Do-it-again
Behavioral: Warning leaflet — The 2-sided color printed A4 leaflet, which systematically covers the most important messages to motivate smoking cessation
  Other Names: Brief leaflet on health warning and smoking cessation
Behavioral: Referral card — The 3-folded "Smoking Cessation Services" card consists of brief information and highlights of existing smoking cessation services, contact methods, motivation information and strong supporting messages or slogans
  Other Names: Smoking Cessation Service Card
Behavioral: COSH booklet — A general smoking cessation self-help booklet
  Other Names: COSH self-help smoking cessation booklet

SUMMARY:
The present study will examine (1) effectiveness of a combined intervention of AWARD advice, active referral, instant messaging and optional cocktail intervention to increase abstinence using a sequential multiple assignment randomised trial (SMART) and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, there are still 615,000 daily cigarette smokers in Hong Kong in 2017 and half will be killed by smoking which accounts for over 7,000 deaths per year. Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP). Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support. Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group.

We propose to use adaptive design for the QTW 2019 specifically a two-phase adaptive design, i.e., a sequential, multiple assignment, randomized trial (SMART) design. Optional cocktail cessation supports will be provided based on smokers' smoking status and preference. The supports, including multimedia messages, active referral plus financial incentive, phone counseling, social support and medications, are empirically evidence-supported and most have been used in our previous QTW interventions.

Therefore, the present study will examine (1) effectiveness of a combined intervention of AWARD advice, active referral, instant messaging and optional cocktail intervention to increase abstinence using a SMART design and (2) explore the use of CBPR model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, a process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3-month
* Able to communicate in Cantonese (including reading Chinese)
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO Smokerlyzer.
* Intent to quit / reduce smoking
* Able to use instant messaging tool (e.g., WhatsApp, WeChat) for communication.

Exclusion Criteria:

* Smokers who have communication barrier (either physically or cognitively)
* Have participation in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Validated abstinence of PIM + OCI vs. RIM + PIM | 6-month follow-up
  PIM + OCI (subgroup A+B+C) vs. RIM + PIM (subgroup D+E+F) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml)
Validated abstinence of OCI vs. RIM in incomplete responders | 6-month follow-up
  OCI (subgroup A) vs. RIM (subgroup E) in incomplete responders (those who are still smoking at 1-month) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml)

SECONDARY OUTCOMES:
Validated abstinence of PIM + OCI vs. RIM + PIM adjusted for potential imbalance of baseline characteristic | 6-month follow-up
  PIM + OCI (subgroup A+B+C) vs. RIM + PIM (subgroup D+E+F) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) adjusted for potential imbalance of baseline characteristic.
Validated abstinence of OCI vs. RIM in incomplete responders adjusted for potential imbalance of baseline characteristic | 6-month follow-up
  OCI (subgroup A) vs. RIM (subgroup E) in incomplete responders (those who are still smoking at 1-month) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) adjusted for potential imbalance of baseline characteristic
Validated and self-reported abstinence of OCI vs. PIM in incomplete responders | 3- and 6-month follow-up
  OCI (subgroup A) vs. PIM (subgroup B) in incomplete responders (those who are still smoking with 1-month) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence
Validated and self-reported abstinence of PIM vs. RIM in incomplete responders | 3- and 6-month follow-up
  PIM (subgroup D) vs. RIM (subgroup E) in incomplete responders (those who are still smoking with 1-month) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence
Validated and self-reported abstinence of PIM vs. RIM | 3- and 6-month follow-up
  PIM (subgroup B+C) vs. RIM (subgroup E+F) on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence
PIM intervention engagement on validated and self-reported abstinence | 3- and 6-month follow-up
  Difference between engagement of PIM intervention vs. no engagement of PIM intervention vs. RIM intervention on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence.
  PIM intervention include subgroup B+C+D, RIM intervention include subgroup E+F.
OCI intervention engagement on validated and self-reported abstinence | 3- and 6-month follow-up
  Difference between engagement of OCI intervention vs. no engagement of OCI intervention vs. engagement of PIM intervention vs. no engagement of PIM intervention vs. RIM intervention on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence.
  OCI intervention include subgroup A, PIM intervention include subgroup B+C+D, RIM intervention include subgroup E+F.
Smoking reduction rate change from baseline at 3- and 6-month follow-up | 3- and 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount
Smoking cessation service use | 3- and 6-month follow-up
  Use of smoking cessation service
Nicotine independence (HSI) on abstinence and intervention engagement | 3- and 6-month follow-up
  Subgroup analyses of high nicotine independence vs. low nicotine independence on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence, and intervention engagement (use of PIM and/or OCI intervention)
Intention to quit analyses on abstinence and intervention engagement | 3- and 6-month follow-up
  Subgroup analyses of high intention to quit vs. low intention to quit on validated abstinence (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) and self-reported abstinence, and intervention engagement (use of OCI intervention and/or PIM intervention and/or RIM intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao SZ, Weng X, Luk TT, Wu Y, Cheung DYT, Li WHC, Tong H, Lai V, Lam TH, Wang MP. Adaptive interventions to optimise the mobile phone-based smoking cessation support: study protocol for a sequential, multiple assignment, randomised trial (SMART). Trials. 2022 Aug 18;23(1):681. doi: 10.1186/s13063-022-06502-7. PMID 35982468